CLINICAL TRIAL: NCT00730860
Title: Treatment of Hepatocellular Carcinoma With Radiofrequency Ablation Associated With Postoperative Transhepatic Arterial Chemoembolization--a Prospective Randomized Clinical Trial
Brief Title: Treatment of Hepatocellular Carcinoma With Radiofrequency Ablation (RFA) Associated With Postoperative TACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, feng xiaobin, Dr Xiaobin Feng, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHB002
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Cancer of Liver
Keywords: radiofrequency ablation; Cancer of Liver; postoperative; transhepatic arterial chemoembolization; prospective
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA+TACE (Experimental): treatment of hepatocellular carcinoma by radiofrequency ablation associated with postoperative transhepatic arterial chemoembolization
  Interventions: Procedure: radiofrequency ablation associated with TACE
- RFA only (Active Comparator): treatment of hepatocellular carcinoma by radiofrequency ablation only
  Interventions: Procedure: radiofrequency ablation only

INTERVENTIONS:
Procedure: radiofrequency ablation associated with TACE — treatment of hepatocellular carcinoma by radiofrequency ablation associated with postoperative transhepatic arterial chemoembolization
  Other Names: Group A
  Arms: RFA+TACE
Procedure: radiofrequency ablation only — treatment of hepatocellular carcinoma by radiofrequency ablation only
  Other Names: Group B
  Arms: RFA only

SUMMARY:
A RCT was conducted to elucidate whether the treatment outcome of HCC could be improved by RFA associated with postoperative TACE.

DETAILED DESCRIPTION:
A randomized study was conducted to elucidate whether the outcome of hepatocellular carcinoma could be improved by radiofrequency ablation associated with postoperative transhepatic arterial chemoembolization.

ELIGIBILITY:
Inclusion Criteria:

* patients with hepatocellular,confirmed by pathological examination
* patients with a live function test showed Child A or B
* Indocyanine green test showed less than 30％ after 15min,and the patients showed a tolerance of RFA and TACE
* Tumor stage is early period(according to Milan Standard),that is,the diameter of single node should be less than 5cm；the node of tumor should be less than 3 and the diameter less than 3cm.
* without metastasis in lymphnode or other organs
* written consent inform assigned

Exclusion Criteria:

* preoperative examination showed malignant thrombosis in the first class branch of portal vein or hepatic vein or vena cava
* metastatic cancer of liver
* patients with a poor tolerance of RFA and TACE
* patients received other therapies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2009-12 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ma Kuansheng, Ph.D, Study Director — Institute of hepatobiliary surgery,Southwest Hospital
Locations (1):
- Institute of hepatobiliary surgery, Chongqing, Chongqing Municipality, China